CLINICAL TRIAL: NCT02542085
Title: Comparison of Hybrid and Laparoscopic Incisional Hernia Repair: A Prospective Randomized Multicentre Study
Brief Title: Comparison of Hybrid and Laparoscopic Incisional Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oulu University Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other); Kymenlaakso Central Hospital Kotka Finland (Other); Päijät Häme Central Hospital (Other); Seinajoki Central Hospital (Other); Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Mirella Ahonen-Siirtola, MD, Oulu University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OuluUH
Record Dates: First submitted 2015-08-31; First posted 2015-09-04 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Incisional Hernia
Keywords: incisional hernia; laparoscopic repair; hybrid repair; seroma; recurrent hernia
MeSH Terms: conditions — Incisional Hernia; Seroma; Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- laparoscopic repair (Active Comparator): patients who are randomized to have a laparoscopic mesh repair
  Interventions: Procedure: Laparoscopic repair
- hybrid repair (Active Comparator): patients who are randomized to have a laparoscopic mesh repair and fascial closure
  Interventions: Procedure: Hybrid repair

INTERVENTIONS:
Procedure: Laparoscopic repair — operative method
  Arms: laparoscopic repair
Procedure: Hybrid repair — operative method
  Arms: hybrid repair

SUMMARY:
Study is a prospective, multicenter, randomized trial evaluating two laparoscopic incisional hernia repair methods: basic laparoscopic mesh repair (lap.) and a hybrid repair (laparoscopic mesh and fascial suturation).

Patients are recruited prospectively from 10 Finnish Hospitals (Oulu, Jorvi, Hyvinkää, Kotka, Seinäjoki, Valkeakoski, Lahti, Kuopio, Kokkola, Loimaa).

Patients are randomized to operative groups (lap. vs hybrid).

Follow-up visits are scheduled at 1- and 12-month after surgery. Patients are evaluated for their clinical status and an ultrasound scan is performed. QoL-questionnaire and pain score (VAS) are reported.

The primary end-points:

* clinically and/or radiologically detected seroma in 1 month control
* clinically and/or radiologically detected recurrent hernia in 1 year control

The secondary end-points:

* peri-and postoperative outcomes/ complications, morbidity, mortality
* duration of hospital stay
* pain scale (VAS)
* Quality of Life (SF/Rand36)

DETAILED DESCRIPTION:
Hypothesis: Using a hybrid method seroma formation and hernia recurrence can be diminished.

Patient exclusion criteria:

Age< 18 y or > 80 y ASA >4 (the American Society of Anaesthesiologists' classification of Physical Health) BMI> 40 A previous mesh repair of the hernia Hernia defect size <2 or >7 cm Emergency operation

Eligible patients are randomized into two operative groups (lap/hybrid). In the laparoscopic group the hernia defect is covered with a Parietex composite mesh (using minimum of 5 cm marginals, Securestrap fixation instrument and four lifting strings. In hybrid group the hernia sack is resected and fascial defect is sutured through a minilaparotomy incision. After this, a mesh repair is performed laparoscopically.

ELIGIBILITY:
Inclusion Criteria:

-Patients with incisional hernia

Exclusion Criteria:

* BMI >40
* ASA IV
* a Prior mesh repair
* Hernia defect size <2 or >7 cm
* Emergency operation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2012-11; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
number of patients with seroma formation | 1 month
number of patients with hernia recurrence | 1 year

SECONDARY OUTCOMES:
number of patients with peri/postoperative complications | up to 1 year
  complications are reported perioperatively, during hospital stay, in 1 month control and in 1 year control
VAS pain scale | 1 year
  Pain scores (VAS) are measured during hospital day (average 3 days), in 1 month control and in 1 year control
Quality of Life | preoperative-1month-1year
  patients are asked to fill SF/rand36-questionnaire preoperatively, in 1 month control and in 1 year control

CONTACTS AND LOCATIONS:
Overall Officials: Tero Rautio, MD, PhD, Study Director — Oulu University Hospital; Mirella Ahonen-Siirtola, MD, Principal Investigator — Oulu University Hospital

REFERENCES:
- [Derived] Ahonen-Siirtola M, Nevala T, Vironen J, Kossi J, Pinta T, Niemelainen S, Keranen U, Ward J, Vento P, Karvonen J, Ohtonen P, Makela J, Rautio T. Laparoscopic versus hybrid approach for treatment of incisional ventral hernia: a prospective randomised multicentre study, 1-year results. Surg Endosc. 2020 Jan;34(1):88-95. doi: 10.1007/s00464-019-06735-9. Epub 2019 Apr 2. PMID 30941550
- [Derived] Ahonen-Siirtola M, Nevala T, Vironen J, Kossi J, Pinta T, Niemelainen S, Keranen U, Ward J, Vento P, Karvonen J, Ohtonen P, Makela J, Rautio T. Laparoscopic versus hybrid approach for treatment of incisional ventral hernia: a prospective randomized multicenter study of 1-month follow-up results. Hernia. 2018 Dec;22(6):1015-1022. doi: 10.1007/s10029-018-1784-2. Epub 2018 Jun 7. PMID 29882170